CLINICAL TRIAL: NCT07086352
Title: Influence of Metastatic Sites on Survival Outcomes and Predictive Factors for Extended Survival in Metastatic Pancreatic Cancer a Retrospective Study
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Dina Gamal Abdelaziz Farrag, residant doctor at assiut university hospital, Assiut University
Other Study IDs: meta site survival pancreatic
Record Dates: First submitted 2025-07-18; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Pancreatic Cancer Metastatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study group: Patients diagnosed with metastatic pancreatic cancer over a defined period (e.g., between 2019 and 2024).
  Study Population: Adult patients (≥18 years) diagnosed with metastatic pancreatic cancer between January 1, 2019, and December 31, 2023.

SUMMARY:
Pancreatic cancer remains one of the most lethal malignancies worldwide, with a 5-year survival rate of less than 10%. The majority of patients are diagnosed at an advanced stage, and nearly 50% present with distant metastases at the time of diagnosis. Despite advances in chemotherapy, such as FOLFIRINOX and gemcitabine-based regimens, the prognosis of metastatic pancreatic cancer (mPC) remains extremely poor, with median overall survival typically ranging between 6 to 11 months.

The pattern of metastasis in pancreatic cancer commonly involves the liver, peritoneum, lungs, and distant lymph nodes. Several studies suggest that the site and extent of metastatic disease may influence survival outcomes, although findings remain inconsistent. For example, liver metastases are frequently associated with worse prognosis, whereas isolated lung metastases may indicate a more indolent disease course. Understanding the prognostic significance of different metastatic sites may provide insight into disease biology and help guide clinical decision-making.

In addition, identifying clinical and pathological factors associated with extended survival could inform treatment stratification, optimize resource allocation, and guide patient counseling. However, limited data exist regarding the predictors of long-term survival in mPC patients, particularly in real-world clinical settings.

Therefore, this retrospective cohort study aims to investigate the influence of metastatic sites on overall survival and to identify potential predictive factors for extended survival among patients with metastatic pancreatic cancer. This information could contribute to more individualized prognostic assessments and potentially support the development of tailored therapeutic strategies.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with metastatic pancreatic cancer over a defined period (e.g., between 2019 and 2024).
* Adult patients (≥18 years) diagnosed with metastatic pancreatic cancer between January 1, 2019, and December 31, 2023.

Exclusion Criteria:

* non metastatic patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with metastatic pancreatic cancer over a defined period (e.g., between 2019 and 2024).
  Study Population: Adult patients (≥18 years) diagnosed with metastatic pancreatic cancer between January 1, 2019, and December 31, 2023.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5 years
  Overall survival (OS) from date of metastatic diagnosis to death or last follow-up.